CLINICAL TRIAL: NCT07329023
Title: An Implementation Science Approach to Evaluating Self-Administered Acupressure for Knee Osteoarthritis in Older-Aged Adults in the Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOIS
Record Dates: First submitted 2025-09-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: knee OA; RCT; pain; osteoarthritis; implementation sciences
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Administered Acupressure (SAA) Intervention for Knee Osteoarthritis Management (Experimental): A training course will be offered to subjects in this group to train them to perform self-acupressure.
  Interventions: Other: Experimental Group: Self-Administered Acupressure (SAA)
- General Health Education (Active Comparator): A booklet of general health education will be offered to the subjects in this group by the research personnel. The research staff will briefly explain the content covered by the booklet and instruct the subjects to read the booklet at home.
  Interventions: Other: Control Group: General Health Education

INTERVENTIONS:
Other: Experimental Group: Self-Administered Acupressure (SAA) — Participants in this group will receive two acupressure training sessions (2 h each, 1 -week apart). The SAA treatment protocol was developed based on TCM meridian theory described in previous studies and modified by the PA and CO-A who is an experienced acupuncturist. The acupoints are indicated for knee pain and are commonly used tested for feasibility in RCT study.
  Participants will be asked to perform the acupressure at home in the morning (within 1 h after waking up) and at night (within 1 h after dinner) every day for 24 weeks. Participants will receive a follow-up phone call from the instructor during the first week to remind them to practice and answer their queries.
  During the intervention and follow-up period, the participants can communicate with the elderly staff/ our research ambassador to ask questions regarding acupressure.
  Other Names: Self-Administered Acupressure(SAA) Intervention for KneeOsteoarthritis Management
  Arms: Self-Administered Acupressure (SAA) Intervention for Knee Osteoarthritis Management
Other: Control Group: General Health Education — The participants of DEC centers in this group will be provided with the general health education booklets despite the same follow-up procedure. The booklets contains general health education information e.g. physical health, sleep health, for the participants' self-reading. The content is based on our previous studies for lifestyle intervention and health information from the government website. They will be told to read the booklet and follow the suggestions in the booklet. They will have the same program after outcome evaluation at 24 weeks.
  Other Names: General Health Education
  Arms: General Health Education

SUMMARY:
This study aims to evaluate the implementation and effectiveness of a self-administered acupressure (SAA) program for knee osteoarthritis (OA) among older adults in Hong Kong community centers. Using a pragmatic cluster randomized controlled trial (RCT) and mixed-methods approach, the research will assess the reach, adoption, implementation, maintenance, and effectiveness of the SAA program in real-world settings, with the goal of informing scalable interventions for knee OA management.

DETAILED DESCRIPTION:
Knee OA is a prevalent and debilitating condition in older adults, often managed with medications that have side effects or nonpharmacological interventions requiring significant behavioral change. Acupressure, a variant of acupuncture, can be self-administered after appropriate training and has shown efficacy in previous RCTs for knee OA. This study will implement the SAA program in district elderly community (DEC) centers across Hong Kong, training frontline workers and older adults to deliver and practice acupressure. The intervention includes two training sessions, ongoing support, and a 24-week follow-up. Effectiveness will be measured by pain reduction, improved knee function, and quality of life, while implementation outcomes will be evaluated using the RE-AIM framework. Qualitative interviews will explore facilitators and barriers to adoption and sustainability.

Objectives:

1. To explore the reach, adoption, implementation, and maintenance of the SAA program among community service units.
2. To examine the effectiveness of the SAA program in relieving pain and improving knee function in middle-aged and older adults in real-world settings.
3. To explore the experiences (facilitators and barriers) of adopting SAA in routine services through qualitative interviews.

Hypothesis

* The SAA program will be effectively implemented in community settings, achieving high reach, adoption, fidelity, and sustainability.
* Participants in the SAA group will experience greater reductions in knee pain and improvements in knee function and quality of life compared to the control group.

Design and subjects:

* Design: Pragmatic cluster randomized controlled trial (RCT) with mixed-methods (quantitative and qualitative).
* Setting: District Elderly Community (DEC) centers in Hong Kong.
* Subjects:

  * Sample Size: 368 older adults (aged ≥60), recruited from DEC centers (8 clusters per group, 23 participants per cluster).
  * Inclusion Criteria: Ethnic Chinese, aged ≥60, able to read Chinese and comprehend Mandarin/Cantonese, probable knee OA (based on clinical criteria), knee pain ≥3 months, pain score ≥3/10, smartphone access, consent.
  * Exclusion Criteria: Medical conditions precluding participation, knee pain from other causes, cognitive impairment, BMI >30, prior knee replacement.

Interventions:

* SAA Group (Focus Group):

  * Two acupressure training sessions (2 hours each, 1 week apart) led by trained instructors.
  * Training includes acupressure technique, knee-health education, practice with feedback, and provision of materials (handouts, rods, logbook).
  * Daily home practice (morning and night) for 24 weeks, with ongoing support via WhatsApp and phone calls.
* General Health Education Group (Control Group):

  * A general health education booklet will be provided during the study period; will receive the SAA program after 24-week outcome evaluation.

Main outcome measures:

The outcome measures will include treatment effectiveness and implementation.

Effectiveness Outcome Primary outcome measure is the numerical rating scale for knee pain. Other measures include Western Ontario and McMaster University Osteoarthritis Index (WOMAC), Short-Form Six-Dimension (SF-6D), Timed Up & Go Test (TUG) and Fast Gait Speed (FGS).

Implementation Outcome RE-AIM framework will be used to evaluate the project, which covers five aspects of reach, effectiveness, adoption, implementation, and maintenance.

Data Analysis

* Quantitative:

  * Double data entry; analysis in SPSS 28.0.
  * Baseline differences controlled as covariates.
  * Linear mixed-effect models to compare changes in primary (NRS pain score) and secondary outcomes (WOMAC, SF-6D, functional tests) over time.
  * Compliance and clinical significance assessed (≥2-point or ≥30% reduction in NRS).
  * Intention-to-treat analysis.
* Qualitative:

  * Thematic content analysis of interview transcripts using NVivo 12.0.
  * Open coding by two independent researchers; themes reviewed for sufficiency and coherence.
* Cost-Effectiveness:

  * QALYs calculated from SF-6D.
  * Incremental cost-effectiveness ratio (ICER) computed.
  * Bootstrapping (5,000 iterations) for uncertainty; cost-effectiveness acceptability curve generated.

ELIGIBILITY:
Inclusion Criteria:

1. ethnic Chinese;
2. aged 60 years or above;
3. able to read Chinese and comprehend Mandarin or Cantonese;
4. fulfilling any 3 of the following criteria. i. morning stiffness 30 min; ii. crepitus on active joint motion; iii. bone tenderness; iv. bone enlargement; or v. no palpable joint warmth (this classification on those with age >50 years yielded 84% sensitivity, and 89% specificity for OA knee diagnosis (25));
5. having knee pain for at least 3 months (26);
6. knee pain 23 on a Likert pain scale from 1-10;
7. having a smartphone (or a family member living together having a smartphone) that is compatible with WhatsApp (based on our previous studies, almost every eligible subject is used to using WhatsApp for social communication); and
8. willing to provide informed consent.

Exclusion Criteria:

1. medical diagnoses or conditions that preclude individuals from active participation (e.g., bleeding disorders, alcohol, or drug abuse);
2. knee pain related to other conditions (cancer, fracture, rheumatoid arthritis, and rheumatism) as screened according to the red flags for further investigation or referral in the NICE 2014 Guidelines for Osteoarthritis of the knee (27);
3. score < 22 in Hong Kong Montreal Cognitive Assessment (HK-MoCA) indicating cognitive impairment that may prevent the understanding of training instructions (28);
4. body mass index over 30, the obese Il criteria for Asians (29) (obese subjects will find great difficulty in performing acupressure on acupoints because physical pressure reaching the muscle is required); and
5. ever had knee-replacement surgery

Further investigation or referral, either at the screening or during the study, will be made whenever necessary.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) for pain severity | Baseline, Week 4, Week 12, Week 24
  Numerical rating scale (NRS) for pain severity The NRS indicates the average pain intensity in the recent one week in the knee. NRS is a single Il-point numeric scale ranging from 0 (no pain) to 10 (greatest pain imaginable). The NRS is a valid and acceptable measure to detect changes in patients' improvement. NRS is chosen as primary outcome because our previous study suggests that the acupressure treatment protocol is more likely to improve global pain intensity. NRS has been used as the primary outcome in recent large-scale RCTs of acupuncture and procedural interventions for knee OA.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index | Baseline, Week 4, Week 12, Week 24
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC): Assesses pain, physical function, and stiffness. A total raw score ranges from 0-96. Scores are often converted to a 0-100 scale (0=best, 100=worst) for standardized reporting, with higher numbers indicating greater disability.
Short Form 6D (SF-6D) | Baseline, Week 4, Week 12, Week 24
  Short Form 6D (SF-6D): Measures quality of life. It is a standard tool used to measure health-related quality of life (HRQoL) by assessing six key areas (physical functioning, role limitations, social functioning, pain, mental health, vitality) from the SF-36. The score ranges from 0 (worst quality of life) to 1 (perfect quality of life).
Timed Up and Go Test | Baseline, Week 4, Week 12, Week 24
  Functional Test: the Timed Up and Go Test to evaluate knee function. It is a assessment of functional mobility and fall risk, especially for older adults, involving timing how long it takes to stand from a chair, walk 3 meters, turn, walk back, and sit down. The time will be recorded (in seconds) for completing the task.
Fast Gait Speed test | Baseline, Week 4, Week 12, Week 24
  Functional Test: Fast Gait Speed test to evaluate knee function. It measures how fast the subject walks by timing them over a 10 m distance where you accelerate for 2m, walk quickly (safely) for 6m , and decelerate for 2m. The time, in seconds, will be recorded for completing the task.
Analgesic Usage | Baseline, Week 4, Week 12, Week 24
  Medication Use:
  Participants may continue their usual medications, with analgesic use recorded during follow-up. They will be asked to fill in a daily log to record their frequency (in times) of analgesic used.
Compliance Assessment | Baseline, Week 4, Week 12, Week 24
  Compliance Assessment:
  Attendance at training and daily practice logged in acupressure logbooks. They are required to fill in their number of practice in the logbook daily.

OTHER OUTCOMES:
Implementation outcome measures -Reach from District Elderly Centers (DEC) | Week 24
  Reach:
  Reached will be evaluated through data documentation, including the screening rate of participants for eligibility
Implementation outcome measures- Adoption | Week 24
  Adoption:
  Adoption will track the number of DEC units that implement the intervention and record reasons for any discontinuation. They will be asked whether their units held any more session of SAA training after our study.
Implementation outcome measures - satisfaction | Week 24
  Implementation:
  Implementation will assess the stakeholders' perception if the intervention is agreeable and the degree to which an intervention is implemented as planned. Satisfaction of participants and providers will be measured using a 15-item questionnaire adapted from a previous community based health-social partnership study, with confirmed validity and reliability. The frontline workers need to record intervention fidelity by using a fidelity checklist for evaluating implementation. The checklist serves to measure the extent to which the core intervention components were delivered as planned. Documentation will be updated by the units with assistance from the research assistant throughout the study period and audited by the research team once every three months.
Implementation outcome measures - Maintenance | Week 24
  The number of SAA program (and participants) launched by the DEC beyond the follow-up period (24-week) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: WIng-Fai YEUNG, Phd, Principal Investigator — School of Nursing. the Hong Kong Polytechnic University, Hong Kong
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
We did not obtain consent from the participants regarding sharing data.